CLINICAL TRIAL: NCT05050032
Title: Study to Assess the Relationship Between Superior Vena Cava Flow and Intraventricular Hemorrhage in Preterm Infants
Brief Title: The Relationship Between Superior Vena Cava Flow and Intraventricular Hemorrhage in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0106381
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Preterm Intraventricular Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The aim of the study was to evaluate the relationship between superior vena cava (SVC) flow measurements within the first 24 hours of life and development of intraventricular hemorrhage in preterm born infants.

DETAILED DESCRIPTION:
A prospective, observational cohort study was carried out on newborns that fulfill the eligibility criteria and delivered at the Alexandria University Maternity Hospital (AUMH).

The Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital with total admissions of approximately 2100 newborn per year of which approximately more than 50% are admitted due to prematurity and its complications.

The study was carried out in 3 phases:

1. First phase: Enrollment and selection phase.
2. Second phase: Monitoring and Evaluation phase.
3. Third phase: Statistical analysis of the data

ELIGIBILITY:
Inclusion Criteria:

* Newborns with very low birth weight (≤1500 g) or ≤ 32 weeks gestation who were admitted to neonatal intensive care unit in the first day of life.

Exclusion Criteria:

* Newborns (more than 32 weeks of gestation
* Newborns with birth weight more than 1500 g.
* Newborns with congenital heart diseases excluding (patent ductus arteriosus and patent foramen ovale)
* Newborns with major congenital malformations.
* Newborns with birth trauma especially basal skull/temporal bone fractures that require hospitalization

Ages: 1 Day to 1 Day | Sex: All
Age Groups: Child
Study Population: Newborns with very low birth weight (≤1500 g) or ≤ 32 weeks gestation who were admitted to neonatal intensive care unit in the first day of life where evaluation of the relationship between superior vena cava (SVC) flow measurements within the first 24 hours of life and development of intraventricular hemorrhage were assessed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Superior vena cava (SVC) flow | Day 1
  This was measured using echocardiography. SVC diameter will be visualized from a high parasternal long axis view. The maximum and minimum internal diameters will be then measured off-line from a frozen two-dimensional image showing the vessel walls at the point where SVC starts to open up into the right atrium. Mean of the maximum and minimum diameter used for the flow calculation.
  * SVC flow velocity will be visualized from a low subcostal view and the pulsed Doppler recording will be made at the junction of the SVC and the right atrium. Velocity time integral (VTI) will be calculated from the Doppler velocity tracings and averaged over 5 consecutive cardiac cycles.
  * SVC flow will be calculated using the method described by Kluckow and Evans:
  SVC flow (ml/kg/min) = {VTI (cm/beat) × 3.14 × (mean SVC diameter2/4) × heart rate (beat/min) }/body weight in kg
Intraventricular hemorrhage (IVH) assessment | Day 1
  Cranial ultrasound will be performed after the echocardiography:
  * Machine: model GE Vivid iq premium.
  * Probe: GE 8C-RS probe with a frequency range of 3.5 - 10 MHz.
  * Cranial ultrasound will be done and any IVH will be noted and classified according to Papile grading:
  Grade I: Hemorrhage limited to germinal matrix Grade II: Blood noted within the ventricular system but not distending it Grade III: Blood in the ventricles with distension of the ventricles Grade IV: Intraventricular hemorrhage with parenchymal extension
Intraventricular hemorrhage (IVH) assessment | Day 3
  Cranial ultrasound will be performed after the echocardiography:
  * Machine: model GE Vivid iq premium.
  * Probe: GE 8C-RS probe with a frequency range of 3.5 - 10 MHz.
  * IVH will be noted and classified according to Papile grading:
  Grade I: Hemorrhage limited to germinal matrix Grade II: Blood noted within the ventricular system but not distending it Grade III: Blood in the ventricles with distension of the ventricles Grade IV: Intraventricular hemorrhage with parenchymal extension
Intraventricular hemorrhage (IVH) assessment | Day 7
  Cranial ultrasound will be performed after the echocardiography:
  * Machine: model GE Vivid iq premium.
  * Probe: GE 8C-RS probe with a frequency range of 3.5 - 10 MHz.
  * Cranial ultrasound will be done and any IVH will be noted and classified according to Papile grading:
  Grade I: Hemorrhage limited to germinal matrix Grade II: Blood noted within the ventricular system but not distending it Grade III: Blood in the ventricles with distension of the ventricles Grade IV: Intraventricular hemorrhage with parenchymal extension
Anterior cerebral artery (ACA) flow velocity assessment | Day 1
  Transcranial Doppler (TCD) ultrasonography was used to assess the anterior cerebral artery flow velocity

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AM Khalifa, MBBCh, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt; Mohamed H Gouda, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Ali M Abd Almohsen, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt; Marwa M Farag, PhD, Study Chair — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt

REFERENCES:
- [Background] Kluckow M, Evans N. Superior vena cava flow in newborn infants: a novel marker of systemic blood flow. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F182-7. doi: 10.1136/fn.82.3.f182. PMID 10794783
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Derived] Farag MM, Gouda MH, Almohsen AMA, Khalifa MA. Intraventricular hemorrhage prediction in premature neonates in the era of hemodynamics monitoring: a prospective cohort study. Eur J Pediatr. 2022 Dec;181(12):4067-4077. doi: 10.1007/s00431-022-04630-5. Epub 2022 Sep 28. PMID 36171508